CLINICAL TRIAL: NCT00231153
Title: A Phase 3, Multicenter, Randomized, Evaluation Committee-Blinded Study to Assess the Efficacy of Topical Omiganan 1% Gel in Preventing Local Catheter Site Infections/Colonization in Patients Undergoing Central Venous Catheterization
Brief Title: Study of Omiganan 1% Gel in Preventing Catheter Infections/Colonization in Patients With Central Venous Catheters
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cadence Pharmaceuticals (Industry)
Responsible Party: Catherine Hardalo, MD. Vice President, Anti Infectives Clinical Development, Cadence Pharmaceuticals, Inc.
Organization: Cadence (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CPI-226-03; EudraCT Number: 2005-003194-24
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Results first posted 2009-08-13 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-06

CONDITIONS: Infection
Keywords: catheter site infection; catheter colonization; catheter related blood stream infection; patients with central venous catheters
MeSH Terms: conditions — Infections | interventions — Omiganan; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Povidone-Iodine 10% (Active Comparator)
  Interventions: Drug: Povidone-Iodine 10%
- omiganan 1% gel (Experimental)
  Interventions: Drug: Omiganan 1% gel

INTERVENTIONS:
Drug: Omiganan 1% gel — Patients randomized to omiganan group will receive an application of omiganan gel around the catheter insertion site following catheter insertion. Every 3 days the dressing will be changed and patients will receive a new application of Omiganan 1% gel.
  Arms: omiganan 1% gel
Drug: Povidone-Iodine 10% — All CVC sites will be disinfected using a 10% povidone-iodine scrub for a minimum of 2 minutes prior to catheter insertion. Patients randomized to the povidone-iodine group will receive no further antiseptic treatment after catheter insertion until dressing changes. Every three days the dressing will be changed and the catheter site will be sterilized with povidone-iodine.
  Arms: Povidone-Iodine 10%

SUMMARY:
The purpose of this study is to determine whether treatment with topical omiganan is more effective than treatment with topical povidone-iodine in preventing local catheter site infections and catheter colonization in patients who have central venous catheters.

DETAILED DESCRIPTION:
Study design:

This is a phase 3, multi-center, randomized, Evaluation Committee-blinded study in patients undergoing noncuffed central venous catheterization using either a single lumen or multi-lumen catheter, and for whom the catheter is expected to be in place for at least 48 hours and for no longer than 28 days. Patients will be randomized within 4 hours of the insertion of the first study CVC.

The first study catheter for all patients must be a noncuffed (nontunneled) central venous catheter (CVC). Additionally, only catheters inserted using povidone iodine to prepare the insertion site are eligible to become study catheters. CVCs will be inserted either into the axillary, jugular, subclavian, or femoral vein. Following the first study CVC insertion, additional CVCs, as well as arterial catheters and PICC lines will be allowed as study catheters. Only catheters that have not been impregnated with an antimicrobial substance (e.g. bonded catheters, antimicrobial impregnated, silver tipped, etc) may be used as study catheters. Study catheters must have a skin/catheter interface; for example, introducers will be allowed as study catheters but any catheter, including a CVC, inserted through the introducer will be deemed a non-study catheter. Once a patient has been randomized to either treatment, all study catheters will receive the same treatment.

NIH (NCID) and/or local hospital guidelines will be followed for maximal sterile barrier precautions. The catheter site will be disinfected using 10% povidone iodine for a minimum of 2 minutes per established CDC guidelines prior to catheter insertion. Patients randomized to the omiganan 1% gel group will receive an application of omiganan 1% gel around the catheter insertion site following catheter insertion. Patients randomized to the povidone iodine group will receive no further antisepsis treatment other than cleansing the site with povidone iodine at dressing changes. For patients in both groups, the catheterization site will be covered with a semitransparent dressing provided by the sponsor.

Every 3 days the dressing will be changed. Skin irritation, erythema and edema will be assessed as well as the presence of purulence, moisture, ecchymosis, abnormally warm tissue temperature and/or site pain/tenderness.

Patients will be discharged from the study following the removal of the final study catheter or on study day 28, whichever is sooner. Patients or their legal representatives will be contacted at least 28 days after study discharge/withdrawal for safety follow-up purposes.

ELIGIBILITY:
Inclusion Criteria:

* New insertion of at least 1 noncuffed (nontunneled) temporary central venous catheter
* Males and females of at least 13 years of age
* A negative urine or serum pregnancy test at baseline

Exclusion Criteria:

* Insertion of, or requirement for, any study catheter impregnated/bonded with an antimicrobial substance
* High probability of death within 14 days of enrollment as assessed by the investigator
* Prior treatment with vancomycin (intravenous administration only), daptomycin, linezolid, or quinupristin/dalfopristin, within 48 hours of first study catheter insertion or prior treatment with tigecycline within one week of first study catheter insertion
* Requirement for topical antibiotic use within 10 cm of any study catheterization site
* Known severe neutropenia (absolute neutrophil count [ANC] < 500 mm3) or recent administration of antineoplastic therapy expected to result in severe neutropenia within 48 hours of first study catheter insertion
* Routine non-complicated coronary artery bypass grafting (CABG) patients, bone marrow transplant (BMT) or solid organ transplant (SOT) patients
* Patients anticipated to be catheterized for less than 48 hours
* Patients who have a suspected or known bloodstream infection at enrollment
* Burn patients or patients with toxic epidermal necrolysis
* Known allergy to adhesive tape or adhesive bandages

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1859 (Actual)
Dates: Start 2005-08; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (57):
- United States (36):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Arcadia, California
  - Glendale, California
  - Long Beach, California
  - Los Angeles, California
  - Madera, California
  - San Diego, California
  - San Francisco, California
  - Torrance, California
  - Denver, Colorado
  - Bridgeport, Connecticut
  - Jacksonville, Florida
  - Miami, Florida
  - Fort Gordon, Georgia
  - Marietta, Georgia
  - Elk Grove Village, Illinois
  - Hoffman Estates, Illinois
  - Louisville, Kentucky
  - Opelousas, Louisiana
  - Shreveport, Louisiana
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - Camden, New Jersey
  - Newark, New Jersey
  - Brooklyn, New York
  - Jamaica, New York
  - Syracuse, New York
  - Oklahoma City, Oklahoma
  - Pittsburgh, Pennsylvania
  - Memphis, Tennessee
  - El Paso, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Lubbock, Texas
  - Morgantown, Virginia
- France (9):
  - Bourg-en-Bresse
  - Brive-la-Gaillarde
  - La Roche-sur-Yon
  - Limoges
  - Montauban
  - Orléans
  - Pau
  - Poitiers
  - Tours
- Germany (4):
  - Halle
  - Jena
  - Leipzig
  - Regensburg
- Spain (8):
  - Alcalá de Henares
  - Barcelona
  - Cadiz
  - El Palmar (Murcia)
  - Las Palmas de Gran Canaria
  - Madrid
  - Palma de Mallorca
  - Seville

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1859 hospitalized patients in the US and EU who required new insertion of short-term central venous catheter were enrolled. Study recruitment began in August 2005 and was completed in April 2008.
Pre-assignment Details: Patients were randomized within 4 hours of insertion of the first study CVC. There were a total of 44 patients who were randomized but never received insertion of CVC or exposure to assigned treatment, who were excluded from the evaluable population and were not reviewed by the Evaluation Committee.
Groups:
- Omiganan 1% Gel: All treated patients: Properly consented patients who received 1 or more doses of omiganan 1% gel with any post baseline observations (Primary Safety Population).
  Modified Intent to Treat Subset: all ITT patients who did not have a BSI at randomization (baseline BSI) as determined by EC adjudication. Patients classified as 'present' (i.e. failure) or 'indeterminate' for baseline BSI were excluded from the MITT population. Patients missing baseline BSI status from EC adjudication were excluded from the MITT population. MITT Among Survivors: patients from the MITT population who did not die on study or who died and were positive (indeterminate or failure)for the study endpoint being analyzed prior to death (as determined by EC adjudication).
- Povidone-Iodine: All treated patients: Properly consented patients who received 1 or more doses of Povidone-Iodine with any post baseline observations (Primary Safety Population).
  Modified Intent to Treat Subset: all ITT patients who did not have a BSI at randomization (baseline BSI) as determined by EC adjudication. Patients classified as 'present' (i.e. failure) or 'indeterminate' for baseline BSI were excluded from the MITT population. Patients missing baseline BSI status from EC adjudication were excluded from the MITT population. MITT Among Survivors: patients from the MITT population who did not die on study or who died and were positive (indeterminate or failure)for the study endpoint being analyzed prior to death (as determined by EC adjudication).
Period: Overall Study
Arm/Group | Omiganan 1% Gel | Povidone-Iodine
Started | 907 (Subjects randomized to omiganan 1% gel who received at least one dose of study treatment.) | 908 (Subjects randomized to povidone-iodine who received at least one dose of study treatment.)
Completed | 690 | 720
Not Completed | 217 | 188

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omiganan 1% Gel | Povidone-Iodine | Total
Number analyzed (Participants) | 907 | 908 | 1815
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 7 | 8
  Between 18 and 65 years | 488 | 499 | 987
  >=65 years | 418 | 402 | 820
Age Continuous [Mean (Standard Deviation); unit: years] | 60.1 (16.82) | 59.4 (17.17) | 59.7 (17.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 350 | 362 | 712
  Male | 557 | 546 | 1103
Region of Enrollment [Number; unit: participants]
  United States | 364 | 366 | 730
  Europe | 543 | 542 | 1085

OUTCOME MEASURES:

1. Primary Outcome: Local Catheter Site Infection (LCSI)
Description: LCSI was defined as a study catheter showing any 2 of the following criteria: erythema >= 2; edema >= 2; presence of purulence, pain, or abnormal study catheter site warmth. In addition, an action must have been taken that indicated a LCSI was present.
Time Frame: study completion
Population: MITT among Survivors: patients from the MITT population (all ITT patients who did not have a baseline BSI) who did not die on study, or who died and were positive (indeterminate or failure) for LCSI prior to death (as determined by EC adjudication).
Measure: Number; unit: Events
Arm/Group | Omiganan 1% Gel | Povidone-Iodine
Number analyzed (Participants) | 793 | 818
Events | 50 | 70
Statistical Analysis 1: Comparison: Omiganan 1% Gel vs Povidone-Iodine; Adequate power was provided to test the null hypothesis that there would be no difference between treatment groups for LCSI. Overall LCSI rate was assumed to be approx. 7.5%, with reduction of LCSI by 40% with omiganan. LCSI rates in placebo and omiganan groups would be 9.375% and 5.625%. Sample size of 1548 in MITT set would provide 80% power to detect this difference between treatments. Sample size was also increased by 19% to account for deaths, for total of 1850 planned patients; Test type: Superiority or Other; p = 0.082, Cochran-Mantel-Haenszel — The primary null hypothesis was tested using the CMH chi-square test stratified region: North America or Europe. Alpha for this test will be 0.05, tow-tailed. No adjustment for multiplicity was performed; Net percentage difference = 2.25, 95% CI [-0.30 to 4.81]

2. Secondary Outcome: Microbiologically-confirmed LCSI
Description: MCLCSI is a subset of EC-adjudicated LCSI for any catheter where there is (1) growth of a recognized pathogen from a culture or any purulence or exudate from the same insertion site, or (2) a positive culture of the subcutaneous segment of the catheter meeting criteria for significant colonization.
Time Frame: study completion
Population: MITT among Survivors: patients from the MITT population (all ITT patients who did not have a baseline BSI) who did not die on study, or who died and were positive (indeterminate or failure) for MCLCSI prior to death (as determined by EC adjudication).
Measure: Number; unit: Events
Arm/Group | Omiganan 1% Gel | Povidone-Iodine
Number analyzed (Participants) | 792 | 818
Events | 31 | 62
Statistical Analysis 1: Comparison: Omiganan 1% Gel vs Povidone-Iodine; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel; Net percentage difference = 3.67, 95% CI [1.40 to 5.93]

3. Secondary Outcome: Catheter Colonization (CC)
Description: CC was defined as a positive culture of any catheter segment >= 15 CFU (roll-plate method) or >999 CFU/ml (sonication method) or a positive blood culture drawn via the catheter where the time-to-positivity difference of catheter line vs. peripheral blood >120 minutes (catheter positive first).
Time Frame: study completion
Population: MITT Among Survivors: patients from the MITT population (all ITT patients who did not have a baseline BSI) who did not die on study, or who died and were positive (indeterminate or failure) for catheter colonization prior to death (as determined EC adjudication).
Measure: Number; unit: Events
Arm/Group | Omiganan 1% Gel | Povidone-Iodine
Number analyzed (Participants) | 845 | 868
Events | 369 | 478
Statistical Analysis 1: Comparison: Omiganan 1% Gel vs Povidone-Iodine; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Net percentage difference = 11.40, 95% CI [6.70 to 16.11]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days